CLINICAL TRIAL: NCT00730288
Title: Safety of ChimeriVax™ Dengue Tetravalent Vaccine in Adult Subjects Previously Immunised With an Investigational Dengue or Yellow Fever Vaccine
Brief Title: Study of ChimeriVax™ Dengue Tetravalent Vaccine in Adult Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CYD10
Record Dates: First submitted 2008-08-06; First posted 2008-08-08 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Dengue; Dengue Fever; Dengue Hemorrhagic Fever; Dengue Virus
Keywords: Dengue; Dengue fever; Dengue hemorrhagic fever; Dengue virus
MeSH Terms: conditions — Dengue; Severe Dengue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Received monovalent Vero dengue vaccine in Study DIV12
  Interventions: Biological: Chimeric dengue serotype (1, 2, 3, 4)
- 2 (Experimental): Received Yellow fever vaccine in Study DIV12
  Interventions: Biological: Chimeric dengue serotype (1, 2, 3, 4)
- 3 (Experimental): Flavivirus-naive subjects
  Interventions: Biological: Chimeric dengue serotype (1, 2, 3, 4)

INTERVENTIONS:
Biological: Chimeric dengue serotype (1, 2, 3, 4) — 0.5 mL, Subcutaneous, 1 dose
  Other Names: ChimeriVax™ Dengue Tetravalent Vaccine
  Arms: 1
Biological: Chimeric dengue serotype (1, 2, 3, 4) — 0.5 mL, Subcutaneous, 1 dose
  Other Names: ChimeriVax™ Dengue Tetravalent Vaccine
  Arms: 2
Biological: Chimeric dengue serotype (1, 2, 3, 4) — 0.5mL, Subcutaneous, 1 dose
  Other Names: ChimeriVax™ Dengue Tetravalent Vaccine
  Arms: 3

SUMMARY:
To evaluate effect of previous flavivirus exposure on the safety and immunogenicity of the ChimeriVax™ dengue tetravalent vaccine

Primary Objectives:

* To describe the safety of one injection of ChimeriVax™ dengue tetravalent vaccine.
* To describe the immune response against dengue before and after one injection of ChimeriVax™ dengue tetravalent vaccine

DETAILED DESCRIPTION:
This study will evaluate a dengue tetravalent vaccine formulation in subjects aged 18 to 40 years and previously immunised with a dengue or YF vaccine.

ELIGIBILITY:
Inclusion Criteria :

* Aged 18 to 40 years on the day of inclusion.
* Informed consent form signed.
* For a woman, inability to bear a child or negative serum pregnancy test.
* Completed the one-year follow-up of Study DIV12.
* Able to attend all scheduled visits and to comply with all trial procedures.
* For a woman of child-bearing potential: use of an effective method of contraception or abstinence for at least four weeks prior to vaccination and at least four weeks after vaccination.

Exclusion Criteria :

* History of thymic pathology (thymoma), thymectomy, or myasthenia gravis.
* Breast-feeding.
* Systemic hypersensitivity to any of the vaccine components or history of a life-threatening reaction to the trial vaccine or a vaccine containing the same substances.
* Previous flavivirus vaccination, e.g. Japanese encephalitis or yellow fever.
* Current abuse of alcohol or drug addiction that may interfere with the subject's ability to comply with trial procedures.
* Planned participation in another clinical trial during the present trial period.
* History of flavivirus infection (confirmed either clinically, serologically or microbiologically).
* Congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding six months, or long-term systemic corticosteroids therapy.
* Chronic illness at a stage that could interfere with trial conduct or completion.
* Blood or blood-derived products received in the past three months.
* Vaccination planned in the four weeks following the trial vaccination.
* Flavivirus vaccination planned during the present trial period.
* Planned travel during the present trial period to areas with high dengue endemicity.
* Subject deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalised without his/her consent.
* Participation in another clinical trial in the four weeks preceding the trial vaccination.
* Any vaccination in the four weeks preceding the trial vaccination.
* Human Immunodeficiency Virus (HIV), Hepatitis B (Ag HBs) or Hepatitis C (HC) seropositivity in blood sample taken at screening.
* Laboratory abnormalities considered clinically significant upon the Investigator's judgement in blood sample taken at screening.
* Positive flavivirus serological test in blood sample taken at screening (for Controls only).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2006-08; Primary Completion 2007-08 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Immunogenicity: To provide information concerning the immunogenicity of ChimeriVax™ | 28, 60 and 180 days post vaccination
Safety: To provide information concerning the safety of ChimeriVax™ | 28 days post-vaccination and entire study duration

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur Inc
Locations (1):
- Adelaide, Australia

REFERENCES:
- [Result] Qiao M, Shaw D, Forrat R, Wartel-Tram A, Lang J. Priming effect of dengue and yellow fever vaccination on the immunogenicity, infectivity, and safety of a tetravalent dengue vaccine in humans. Am J Trop Med Hyg. 2011 Oct;85(4):724-31. doi: 10.4269/ajtmh.2011.10-0436. PMID 21976579